CLINICAL TRIAL: NCT06052254
Title: A Double-Blind, Placebo-Controlled Evaluation of the Dexmedetomidine Transdermal Systems for Agitation Associated With Dementia of the Alzheimer's Type
Brief Title: Dexmedetomidine Transdermal Systems (DMTS) Treatment for Agitation Associated With Dementia of the Alzheimer's Type
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teikoku Pharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPU-DMT-02-2213
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Agitation
Keywords: Agitation; Dementia; DMTS
MeSH Terms: conditions — Psychomotor Agitation; Dementia

STUDY DESIGN:
Intervention Model Description: Subjects in each treatment group will receive a total of 4 patches/systems during the study (2 patches/system each dosing period).
  For the second dosing period, subjects will receive the same treatment administered as the first dosing period. An independent data monitoring committee will periodically review safety data to confirm the safety/tolerability of the dose. Subjects will reside in their care facility for the duration of the trial. The following assessments will be performed: agitation assessments (frequency and severity); sedation-level assessments; safety assessments (vital signs including oxygen saturation by pulse oximetry (SpO2)); DMTS/matching placebo adhesion assessments; and skin irritation assessments. In addition, blood samples will be collected for determination of plasma concentrations of dexmedetomidine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sponsor, the investigator, personnel at the clinical study unit who are directly involved with monitoring and/or performing study procedures and assessments, and the subjects will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 12 cm2 - 2 Active DMTS Patches (Active Comparator): 2 Active DMTS patches will be applied to the upper back and worn for 4 days (96 hours) followed 14 days later with the same treatment for an additional 4-day treatment for subjects that are eligible for a second dosing.
  Interventions: Drug: 12 cm2 - 2 Active DMTS Patches
- 6 cm2 - 1 Active and 1 Placebo DMTS Patches (Active Comparator): 1 Active and 1 Placebo DMTS patches will be applied to the upper back and worn for 4 days (96 hours) followed 14 days later with the same treatment for an additional 4-day treatment period for subjects that are eligible for a second dosing.
  Interventions: Drug: 6 cm2 - 1 Active and 1 Placebo DMTS Patches
- Placebo - 2 Placebo DMTS Patches (Placebo Comparator): 2 Placebo DMTS patches will be applied to the upper back and worn for 4 days (96 hours) followed 14 days later with the same treatment for an additional 4-day treatment period for subjects that are eligible for a second dosing.
  Interventions: Drug: Placebo - 2 Placebo DMTS Patches

INTERVENTIONS:
Drug: 12 cm2 - 2 Active DMTS Patches — 2 Active DMTS patches applied to the upper back followed 14 days later by another application of 2 Active DMTS patches. Each application will be worn for 4 days (96 hours)
  Arms: 12 cm2 - 2 Active DMTS Patches
Drug: 6 cm2 - 1 Active and 1 Placebo DMTS Patches — 1 Active and 1 Placebo DMTS patches applied to the upper back followed 14 days later by another application of 1 Active and 1 Placebo DMTS patches. Each application will be worn for 4 days (96 hours)
  Arms: 6 cm2 - 1 Active and 1 Placebo DMTS Patches
Drug: Placebo - 2 Placebo DMTS Patches — 2 Placebo DMTS patches applied to the upper back followed 14 days later by another application of 2 Placebo DMTS patches. Each application will be worn for 4 days (96 hours)
  Arms: Placebo - 2 Placebo DMTS Patches

SUMMARY:
The primary objective of this study is to evaluate the efficacy of DMTS on frequency and severity of agitation associated with dementia of the Alzheimer's type, compared with placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, two application study of DMTS or matching placebo over a 4-day treatment period, followed 14 days later with the same treatment (active or placebo) for an additional 4-day treatment period for subjects that are eligible for second dosing.

Eligible subjects will be screened up to 21 days prior to study start.

Eligible subjects will be randomized 1:1:1 to treatment with 1 DMTS and 1 matching placebo, 2 DMTS, or 2 matching placebos.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent (subject or legally authorized representative [LAR]).
2. Male or female, residing in a care facility.
3. Has a diagnosis of dementia of probable Alzheimer's Disease (AD) based on National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria (2018). The clinical diagnosis of "probable Alzheimer's Disease (AD)" will be based on the 2018 National Institute on Aging-Alzheimer's Association (NIA-AA) diagnostic criteria, which includes patient biomarker data as part of the research diagnosis (Jack et al., 2018). If patient biomarker data are unavailable, per the 2018 NIA-AA diagnostic criteria, the clinical diagnosis of probable AD will be based on the 2011 NIA-AA criteria (McKhann et al., 2011).
4. Had two or more episodes (using a 7-day lookback period) of agitation that impairs social activities, requires staff or medical intervention, or impairs ability for functional activities of daily living at Screening.
5. Had an ABS total score ≥ 22 at least once during Day -4 to Day -1 when assessing eligibility on Day 1 Pre-randomization.
6. Has gone a minimum of 1 week with no change in medication prior to Screening.
7. Has a score of ≤ 23 on the Mini-Mental State Examination (MMSE) at Screening.
8. Female subjects who are:

   1. Not pregnant, not lactating, and not planning to become pregnant during the study or for 1 menstrual cycle thereafter and
   2. Surgically sterile; or postmenopausal (ie, amenorrhea for ≥2 years as reported by subject/caregiver; postmenopausal status will be confirmed with FSH test); or have a monogamous partner who is surgically sterile; or have a same gender sex partner; or is using double-barrier contraception; or practicing abstinence; or using an insertable, injectable, transdermal, or combination oral contraceptive for 3 months prior to the study, during the study, and for 1 month following the study.
9. Male subjects who have female sex partners of childbearing potential must be surgically sterile or commit to use a reliable method of birth control during the study and for 1 month following the study. Reliable contraception is defined as: A tubal ligation, condom with spermicidal gel, an approved hormonal contraceptive such as oral contraceptives, emergency contraception used as directed, patches, implants, injections, rings, or hormone releasing or copper intrauterine device (IUD).
10. Has a body weight > 50 kg, and body mass index of 20 to 38 kg/m2, inclusive.
11. Subject or LAR able to understand the study procedures, comply with all study procedures, and agree to participate in the study program for its full duration.
12. Has lived in facility for at least 7 days prior to screening and will remain in facility through the completion of Follow-Up assessments.

Exclusion Criteria:

1. Has a known sensitivity to dexmedetomidine or any excipient in the DMTS/placebo.
2. Has a skin abnormality (eg, scar, tattoo) or unhealthy skin condition (eg, burns, wounds) at the DMTS/matching placebo application site, according to examination by the investigator at screening.
3. Has a clinically significant abnormal clinical laboratory test value as determined by the investigator.
4. Has agitation caused by acute intoxication.
5. Has significant risk of suicide or homicide per investigator's assessment, or any patient with an answer of "yes" to Items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS).
6. Has a history of or positive test results for the human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
7. Has a clinically significant history or clinically significant manifestation of any of the following, as determined by the investigator: a renal (including an estimated glomerular filtration rate [eGFR] below the appropriate age- and gender-specific range [see Section 8.1.3.2]), hepatic (including any evidence of ascites and/or a Child-Pugh hepatic impairment score > 6 [Appendix G]), cardiovascular, metabolic, neurologic, or psychiatric condition; congestive heart failure, peptic ulcer, gastrointestinal bleeding, or other condition that may preclude participation in the study.
8. Has a history of physician-diagnosed migraine, frequent non-vascular headaches (> 5 per month), seizures, or are currently taking anticonvulsants.
9. Has a history of syncope or other syncopal attacks.
10. Has present and/or significant history of postural hypotension (determined through examination by the investigator or designee) or history of severe dizziness or fainting on standing in the opinion of the investigator.
11. Has evidence of a clinically significant 12-lead ECG abnormality.
12. Has an average heart rate < 60 or > 100 bpm, systolic blood pressure (BP) < 90 or > 140 mmHg, or diastolic BP < 60 or > 90 mmHg, measured in 3 sequential positions (supine after 5 minutes; sitting after 1 minute; and standing after 2 minutes) and after the sequence has been completed 3 times.
13. Has a history of alcohol abuse or prescription/illicit drug abuse within the previous 5 years.
14. Has positive results on the urine drug screen or alcohol breath test indicative of drugs of abuse or alcohol use at screening.
15. Is receiving concurrent therapy that can interfere with the evaluation of efficacy or safety, such as any drug that in the investigator's opinion may exert significant synergistic interactions with dexmedetomidine.

    Medications with potential cardiac effects (eg, hypotension, bradycardia) and medications that may cause sedation (such as quetiapine [Seroquel®]), are permissible if the subject has been on a stable dose for a minimum of 30 days prior to Screening and the investigator deems it appropriate.

    Medications given for the treatment of chronic agitation are permissible if the subject has been on a stable dose for a minimum of 30 days prior to Screening.
16. Uses any natural health products (including chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian, and excluding vitamins or mineral supplements) within 7 days prior to study drug administration and throughout the study, unless in the opinion of the investigator or designee the product will not interfere with the study procedures or data integrity or compromise the safety of the subject.
17. Had symptoms of an upper respiratory tract infection within 7 days prior to dosing of the study drug.
18. Utilized oral or injectable corticosteroids within 7 days prior to dosing of the study drug (intranasal and topical corticosteroid use during this time period is allowed).
19. Received any investigational product within 30 days prior to dosing of the study drug.
20. Received DMTS in a previous clinical trial.
21. Has a Johns Hopkins Fall Risk Assessment Score of > 13.
22. In the opinion of the investigator or designee, is considered unsuitable for study entry and/or is unlikely to comply with the study protocol for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Agitated Behavior Scale (ABS) total score from baseline (Day -4 to Day -1 mean score) to the 96 hours of first application (Day 1 to Day 4). | Baseline (Day -4 to Day -1) to 96 hours after first application (Day 1 to Day 4)
  The ABS [5] is a 14-item scale developed to allow objective assessment of agitated behavior, particularly serial assessments for the evaluation of interventions to reduce agitation. The ABS Total Score ranges from 14 to 56. A total score of 21 or less is considered Normal; 22 to 28 is considered Mild; 29 to 35 Moderate; and 36 or more Severe Agitation.

SECONDARY OUTCOMES:
Change in Clinical Global Impression Scale - Severity (CGI-S) score at 96 hours post-application (Day 5) relative to Pre-randomization (Day 1) baseline. | Day1 (Pre-randomization), Day 5
  The CGI-S is a one item, 4-point (1-4) clinician-rated scale in which higher ratings indicate greater severity of agitation.
Change in ABS total score from baseline (Day -4 to Day -1 mean score) to the 168 hours post first application (Day 1 to Day 7). | From Day -4 through Day 7
  The ABS [5] is a 14-item scale developed to allow objective assessment of agitated behavior, particularly serial assessments for the evaluation of interventions to reduce agitation.
Change in CGI-S score at 168 hours post application (Day 8) relative to Day 1 Pre-randomization baseline. | Day1 (Pre-randomization), Day 8
  The CGI-S is a one item, 4-point (1-4) clinician-rated scale in which higher ratings indicate greater severity of agitation.
Percentage of subjects meeting the criteria for Day 15 DMTS/placebo application. | Day 15
  Number of subjects that meet the criteria for Day 15 dosing.
Change from Pre-randomization Day 1 baseline score (Day -7 to Day -1 lookback) to 168 hours post application score (Day 1 to Day 7 lookback) in the Neuropsychiatric Inventory - Nursing Home Version (NPI-NH). | Day -7, Day 7
  The NPI-NH assesses the severity and frequency of each neuropsychiatric symptom and the amount of caregiver/study partner distress engendered by each of the neuropsychiatric symptoms based on a series of scripted questions administered to a designated informant with a 7-day lookback period. The frequency scale uses a 4-point scale (1-4), and the severity uses a 3-point scale (1-3) with the higher score indicating more frequency or severity.

CONTACTS AND LOCATIONS:
Overall Officials: James Song, MS, Study Director — Teikoku Pharma USA, Inc.
Locations (3):
- United States (3):
  - Elixia MA, LLC, Springfield, Massachusetts
  - Vitalix, Worcester, Massachusetts
  - BioBehavioral Health, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No